CLINICAL TRIAL: NCT03134820
Title: Time of Treatment With Low Molecular Weight Heparins in Cancer Patients With Thromboembolic Disease. Procoagulant Role of Phospholipid-dependent Microparticles.
Brief Title: Time of Treatment With LMWH in Cancer Patients With Thromboembolic Disease
Status: Completed | Type: Observational
Sponsor: Delos Clinical (Other)
Responsible Party: Principal Investigator, Remedios Otero Candelera, MD Ph D, Hospitales Universitarios Virgen del Rocío
Other Study IDs: Hispalis study
Record Dates: First submitted 2017-04-26; First posted 2017-05-01 (Actual); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Venous Thromboembolism; Pulmonary Thromboembolisms; Cancer
Keywords: Low molecular weight heparins; Procoagulants; Phospholipid-dependent Microparticles
MeSH Terms: conditions — Venous Thromboembolism; Pulmonary Embolism; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cancer is the most important acquired risk factor of thromboembolisms. More than 20% of all episodes of venous thromboembolism (VT) or pulmonary thromboembolisms (PT) are cancer related. Cancer patients with VT or PT are treated with low molecular weight heparins (LMWH) during at least 3 months, but nowadays the duration of treatment is not accurately determined.

The D-Dimer determination has been used like recurrence predictors after LMWH treatment suspension, but in cancer patients the useful is limited. Phospholipid-dependent microparticles could been used like recurrence predictors in cancer patients and tailored the duration of LMWH treatment for each patient.

DETAILED DESCRIPTION:
We are carrying out a study in Cancer-associated-thromboembolism patients in order to decide the suitable anticoagulation time. A set of exclusion criteria is being used to determine in which patients LMWH will be withdrawn. Patients are being followed after LMWH withdrawal until 6 months. Blood samples are being taken at baseline (LMWH withdrawal), 3 weeks and 3 months after. We will look for association between several biomarkers and venous thromboembolism recurrences.

ELIGIBILITY:
Inclusion Criteria:

* Patient with diagnosis of cancer (any) and diagnosis of pulmonary thromboembolism (PT) or venous thromboembolism (VT) , in treatment with low molecular weight heparin (LMWH).
* Patients treated with LMWH since cancer diagnostic.
* Signed informed consent sheet

Exclusion Criteria:

* Patients with life expectancy lower than 6 months
* Pregnancy woman
* Patients with cerebral metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with diagnosis of cancer (any) and diagnosis of pulmonary thromboembolism (PT) or venous thromboembolism (VT) , in treatment with low molecular weight heparin (LMWH).
Sampling Method: Non-Probability Sample
Enrollment: 352 (Actual)
Dates: Start 2015-12-15 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Recurrence thromboembolisms | 3 months
  Venous thromboembolisms or Pulmonary thromboembolism recurrence after LMWH suppression
Recurrence thromboembolisms | 6 months
  Venous thromboembolisms or Pulmonary thromboembolism recurrence after LMWH suppression

SECONDARY OUTCOMES:
Hemorrhagic events | 6 months
  Hemorrhagic events due to LMWH treatment
Thromboembolic event attributable death | 6 months
  Death related to embolic event

CONTACTS AND LOCATIONS:
Overall Officials: Remedios Otero Candelera, MD PhD, Study Chair — Hospital Universitario Virgen del Rocío IBIS; Teresa Elias, MD PhD, Principal Investigator — Hospitales Universitarios Virgen del Rocío; Isabel Blasco, MD, Principal Investigator — Hospital Universitario Virgen Macarena; Maria Rodriguez, MD, Principal Investigator — Hospital Universitario de Valme

IPD SHARING:
Plan to Share IPD: No